CLINICAL TRIAL: NCT02911896
Title: Physical Function in Critical Care (PaciFIC): An Multi-centre Observational Study
Brief Title: Physical Function in Critical Care (PaciFIC)
Acronym: PaciFIC
Status: Completed | Type: Observational
Sponsor: University of Melbourne (Other)
Collaborators: Melbourne Health (Other); Flinders Medical Centre (Other Government); National University Hospital, Singapore (Other); Escola Superior da Saude, Brazil (Unknown)
Responsible Party: Principal Investigator, Selina M Parry, Dr, PhD, Grad Cert Uni Teaching, B.Physio (Hons), University of Melbourne
Other Study IDs: 2015026
Record Dates: First submitted 2016-07-25; First posted 2016-09-22 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Intensive Care (ICU) Myopathy
Keywords: physical function; critical care
MeSH Terms: conditions — Muscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Impairment in physical function is a significant problem for survivors of critical illness. There is a growing urgency to develop a core set of outcome measures, which can be adopted in clinical and research practice to evaluate efficacy in response to interventions such as rehabilitation.

Phase 1: Development of a new outcome measure. This study aims to examine the development of a single outcome measure which may be able to be utilised across the continuum of recovery of critical illness in the evaluation of physical function. The study will involve examination of two common physical function measures - the Physical Function in intensive care test scored (PFIT-s) and De Morton Mobility Index (DEMMI) and the development of a new measure based on rasch principles which may be able to capture physical functioning changes in individuals with critical illness. Aims: (1) To determine the clinical utility of two physical function measures (DEMMI and PFIT-s) when used in isolation across the hospital admission; and (2) To transform the (15-item) DEMMI and (4-item) PFIT-s into a single measure to evaluate function in intensive care survivors using Rasch analytical principles.

Phase 2: Measurement properties of the PACIFIC physical function outcome measure in an independent validation sample.

DETAILED DESCRIPTION:
Consecutive eligible patients will be recruited into the study.

Phase 1: Two outcome measures - PFIT-s and DEMMI will be performed within 24 hour period. Order of testing will be randomised to minimise testing bias. Time-points of assessment are: awakening, ICU discharge and hospital discharge. Weekly measures will also be performed if required in ICU and/or ward settings for up to a maximum of 30 days in each setting. The measurement properties of the individual tools PFIT-s and DEMMI will be examined (e.g. validity, responsiveness).

Phase 2: Based on the findings in Phase 1 a new single outcome measure will be developed. In the second phase examination of the measurement properties of the tool will be undertaken including (reliability, validity, responsiveness).

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years of age
* Mechanically ventilated > 48 hours
* Premorbid able to ambulate at least 10m independently prior to ICU admission (+/- gait aid)

Exclusion Criteria:

* Premorbid physical or cognitive impairment which would prevent ability to perform functional measures
* New neurological impairment such as stroke or spinal cord injury
* Trauma or orthopaedic injury requiring period of immobilization or non weight bearing status
* Traumatic brain injury with focal neurology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multi-centre study conducted in four acute hospitals: Royal Melbourne Hospital, Melbourne, Australia; Flinders Medical Centre, Adelaide, Australia; Escola Superior da Saude, Brasilia, Brazil; and National University Hospital, Singapore.
Sampling Method: Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2015-08; Primary Completion 2016-12 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change in Physical Function in Intensive Care Test scored (PFIT-s) and De Morton Mobility Index from ICU awakening to hospital discharge | Baseline to hospital discharge (up to 3 months)
  Both measures are primary - there will be a single measure developed as composite in line with aims of this observational study

CONTACTS AND LOCATIONS:
Overall Officials: Dr Selina M Parry, PhD, Principal Investigator — University of Melbourne
Locations (4):
- Australia (2):
  - University of South Australia and Flinders Medical Centre, Adelaide, South Australia
  - Royal Melbourne Hospital, Melbourne, Victoria
- Escola superior de ciências da saúde ESCS, Brazil, Brazil
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Parry SM, Granger CL, Berney S, Jones J, Beach L, El-Ansary D, Koopman R, Denehy L. Assessment of impairment and activity limitations in the critically ill: a systematic review of measurement instruments and their clinimetric properties. Intensive Care Med. 2015 May;41(5):744-62. doi: 10.1007/s00134-015-3672-x. Epub 2015 Feb 5. PMID 25652888
- [Result] Parry SM, Denehy L, Beach LJ, Berney S, Williamson HC, Granger CL. Functional outcomes in ICU - what should we be using? - an observational study. Crit Care. 2015 Mar 29;19(1):127. doi: 10.1186/s13054-015-0829-5. PMID 25888469